CLINICAL TRIAL: NCT01467271
Title: Observational Study on the Incidence of NSF in Renal Impaired Patients Following Dotarem Administration
Acronym: NSsaFe
Status: Completed | Type: Observational
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: DGD-55-003
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-09

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose of this study is to prospectively estimate the incidence of Nephrogenic Systemic Fibrosis (NSF) in patients with moderate to severe renal impairment after administration of Dotarem®

DETAILED DESCRIPTION:
All patients will be followed up during 2 years after Dotarem® administration to collect data on any suspected NSF or NSF-related symptoms

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe and end stage renal impairment or dialysis, scheduled for a contrast-enhanced Magnetic Resonance Imaging (MRI) with Dotarem

Exclusion Criteria:

* Patient who has received a Gadolinium Based Contrast Agent (GBCA) within the past 12 months prior to inclusion in this study except if the GBCA received is Dotarem

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with moderate to severe and end stage renal impairment or dialysis
  * Patients scheduled for a contrast-enhanced MRI with Dotarem
Sampling Method: Non-Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Desché, MD, Study Director — Guerbet
Locations (27):
- United States (4):
  - Covenant Health Care, Saginaw, Michigan
  - St. Louis University Medical Center, St Louis, Missouri
  - Abington Memorial Hospital, Philadelphia, Pennsylvania
  - University of Texas Health Science Center, San Antonio, Texas
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Belgium (3):
  - UZ Brussel, Brussels
  - AZ St Lucas, Ghent
  - H. Hartziekenhuis, Roeselare
- Colombia (2):
  - Hospital Universitario de San Ignacio, Bogotá
  - IATM (Instituto de alta tecnologia Medica de Antoquia), Medellín
- France (2):
  - Hôpital Necker - Enfants malades, Paris
  - Hôpital Bois-Guillaume - CHU de Rouen, Rouen
- Germany (2):
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Institute of Radiology and Neuroradiology, Frankfurt
- Italy (3):
  - Instituto Tumori Pascale, Napoli
  - Ospedale Santa Maria, Pozzuoli
  - Universita campus Biomedico, Roma
- South Korea (4):
  - Soonchunhyang Univ. Bucheon Hospital, Gyeonggi-do
  - Uijeongbu St. Mary's Hospital, Gyeonggi-do
  - Chung-Ang Univ. Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
- Spain (2):
  - Hospital Clínico San Carlos de Madrid, Madrid
  - CRC Hospital Universitari Sant Joan de Reus, Reus
- Turkey (Türkiye) (2):
  - Dişkapi Etlik Polikliniği, Ankara
  - Medeniyet University Goztepe Research and Training Hospital, Istanbul
- United Kingdom (2):
  - Royal Liverpool University Hospital, Liverpool
  - University Hospital of North Staffodshire, Stoke-on-Trent

RESULTS

PARTICIPANT FLOW:
Groups:
- All Included Patients: All patients included in the study.
Period: Overall Study
Arm/Group | All Included Patients
Started | 540
Completed | 338
Not Completed | 202
Not completed — Death | 84
Not completed — Lost to Follow-up | 83
Not completed — Retraction of patient's consent | 21
Not completed — Other reason | 14

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: The safety population included all patients receiving at least one injection of contrast media regardless of the quantity.
Arm/Group | Safety Population
Number analyzed (Participants) | 539
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224
  Male | 315
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Colombia | 15
  South Korea | 117
  Argentina | 2
  Turkey | 50
  Belgium | 121
  United States | 76
  Italy | 37
  United Kingdom | 9
  France | 23
  Germany | 77
  Spain | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Moderate to Severe Renal Impairment Who Develop Nephrogenic Systemic Fibrosis (NSF) After Administration of Dotarem
Time Frame: All patients were followed up during 2 years after Dotarem administration.
Measure: Count of Participants; unit: Participants
Groups:
- NSF Population: The NSF population included patients with the NSF follow-up questionnaire completed.
Arm/Group | NSF Population
Number analyzed (Participants) | 446
Participants | 0

ADVERSE EVENTS:
Time Frame: The collection of adverse events was done during the MRI examination and during the usual follow-up post-contrast agent administration (mainly less than 30 minutes post-injection).
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/539
Serious Adverse Events (participants affected / at risk) | 0/539
Other Adverse Events (participants affected / at risk) | 0/539

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2012-07-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT01467271/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT01467271/SAP_001.pdf